CLINICAL TRIAL: NCT01866033
Title: An Open-Label, Sequential and 2-Way Crossover Pharmacokinetic Study to Assess the Absolute Bioavailability of Oral PCI-32765 and the Effect of Grapefruit Juice on the Bioavailability of PCI-32765 in Healthy Subjects
Brief Title: A Study to Assess the Absolute Bioavailability of Oral PCI-32765 and the Effect of Grapefruit Juice on the Bioavailability of PCI-32765 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR101359; PCI-32765CLL1011 (Other: Janssen Research & Development, LLC); 2013-000963-96 (EudraCT Number)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Volunteer
Keywords: Healthy volunteer; PCI-32765; PCI 45227; 13C6 PCI-32765; Pharmacokinetic; Bioavailability
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PCI-32765 (Experimental): During Period 1, all patients will receive PCI-32765 560 mg administered by mouth (Treatment A). In Periods 2 and 3, patients will receive PCI-32765 560 mg administered by mouth without grapefruit juice (Treatment B) and PCI-32765 140 mg administered by mouth with grapefruit juice (Treatment C) according to a randomization schedule. An intravenous dose of 13C6 PCI-32765 will be administered 2 hours after each oral dose for reference purposes.
  Interventions: Drug: PCI-32765 (Treatment A); Drug: PCI-32765 (Treatment B); Drug: PCI-32765 (Treatment C); Drug: 13C6 PCI-32765 (reference)

INTERVENTIONS:
Drug: PCI-32765 (Treatment A) — 560 mg capsules administered by mouth on Day 1, Period 1
Drug: PCI-32765 (Treatment B) — 560 mg capsules administered by mouth (without grapefruit juice) on Day 1 during Period 2 or 3 according to randomization schedule
Drug: PCI-32765 (Treatment C) — 140 mg capsule administered by mouth (with grapefruit juice) on Day 1 during Period 2 or 3 according to randomization schedule
Drug: 13C6 PCI-32765 (reference) — 100 mcg administered intravenously 2 h after study drug

SUMMARY:
The purpose of this study is to assess the absolute bioavailability of oral PCI-32765 and the effect of grapefruit juice on the absorption of PCI-32765 in healthy adult participants.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known), sequential and 2-way crossover design, pharmacokinetic (study of what the body does to a drug) study to assess the absolute bioavailability of oral (by mouth) PCI-32765 and the effect of grapefruit juice on the absorption of PCI-32765 in approximately 8 healthy adult participants. The duration of the study is approximately 45 days (screening, treatment, and follow-up). All patients will receive PCI-32765 560 mg (Treatment A) administered by mouth in the first period and Treatment B (560 mg administered by mouth without grapefruit juice) and Treatment C (140 mg administered by mouth with grapefruit juice) according to a randomization schedule in Periods 2 and 3. Participants will fast overnight for at least 10 hours prior to study drug dosing. Participants will stay in the study center for pharmacokinetic sampling. Serial pharmacokinetic samples will be collected before dosing and over 72 hours after dosing and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Women must be postmenopausal or surgically sterile
* Men must agree to use an adequate contraception method during the study and for 3 months after receiving the last dose of study drug, and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Body mass index between 18 and 30 kg/m2 and body weight not less than 50 kg
* Blood pressure (after lying down for 5 minutes) between 90 and 140 mmHg systolic and no higher than 90 mmHg diastolic

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, history of immune disorders (eg, lupus, rheumatoid arthritis, psoriatic arthritis), or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, coagulation, PFA 100, clinical chemistry, or urinalysis at screening
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram at screening
* Use of aspirin, NSAIDs, thienopyridines, vitamin E supplements, fish oil, or flax seed within 1 week before PFA-100 assay test at screening
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol, hormonal replacement therapy and topical anesthetics (intravenous administration), within 14 days before the first dose of the study drug is scheduled
* Use of herbal supplements within 30 days of the first dose administration
* History of drug or alcohol abuse according to the Diagnostic and Statistical Manual of Mental Disorders (4th edition) (DSM-IV) criteria within 2 years before screening or positive test result(s) for alcohol and/or drugs of abuse at screening and Day -1 of each treatment period
* History of clinically significant allergies, especially known hypersensitivity or intolerance to sulfonamide or beta-lactam antibiotics
* Known allergy to the study drug or any of the excipients of the formulation
* Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study
* Received an experimental drug or used an experimental medical device within 1 month or within a period less than 10 times the drug's half life, whichever is longer, before the first dose of the study drug is scheduled
* Unable to swallow solid, oral dosage forms whole with the aid of water
* If a woman, pregnant, breast-feeding or planning to become pregnant during the study
* Positive test for human immunodeficiency virus 1 and 2 antibodies, hepatitis B surface antigen, or hepatitis C antibodies
* History of smoking or use of nicotine-containing substances within the previous 2 months or positive cotinine test
* Preplanned surgery or procedures that would interfere with the conduct of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to 24 hours of PCI-32765 | Predose, and postdose at 30 min, 1 h, 1.5 h, 2 h, 2 h 2 min, 2 h 5 min, 2.2 h, 2.25 h, 2.5 h, 3 h, 3.5 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h, 72 h
Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration of PCI-32765 | Predose, and postdose at 30 min, 1 h, 1.5 h, 2 h, 2 h 2 min, 2 h 5 min, 2.2 h, 2.25 h, 2.5 h, 3 h, 3.5 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h, 72 h
Area under the plasma concentration-time curve from time 0 to infinite time of PCI-32765 | Predose, and postdose at 30 min, 1 h, 1.5 h, 2 h, 2 h 2 min, 2 h 5 min, 2.2 h, 2.25 h, 2.5 h, 3 h, 3.5 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h, 72 h
Absolute bioavailability of PCI-32765 | Predose, and postdose at 30 min, 1 h, 1.5 h, 2 h, 2 h 2 min, 2 h 5 min, 2.2 h, 2.25 h, 2.5 h, 3 h, 3.5 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h, 72 h

SECONDARY OUTCOMES:
Maximum observed plasma concentration of PCI-32765 | Predose, and postdose at 30 min, 1 h, 1.5 h, 2 h, 2 h 2 min, 2 h 5 min, 2.2 h, 2.25 h, 2.5 h, 3 h, 3.5 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h, 72 h
Time to reach the maximum plasma concentration of PCI-32765 | Predose, and postdose at 30 min, 1 h, 1.5 h, 2 h, 2 h 2 min, 2 h 5 min, 2.2 h, 2.25 h, 2.5 h, 3 h, 3.5 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h, 72 h
Elimination half-life of PCI-32765 | Predose, and postdose at 30 min, 1 h, 1.5 h, 2 h, 2 h 2 min, 2 h 5 min, 2.2 h, 2.25 h, 2.5 h, 3 h, 3.5 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 36 h, 48 h, 72 h
Number of participants affected by an adverse event | Up to 30 days after the last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] de Jong J, Sukbuntherng J, Skee D, Murphy J, O'Brien S, Byrd JC, James D, Hellemans P, Loury DJ, Jiao J, Chauhan V, Mannaert E. The effect of food on the pharmacokinetics of oral ibrutinib in healthy participants and patients with chronic lymphocytic leukemia. Cancer Chemother Pharmacol. 2015 May;75(5):907-16. doi: 10.1007/s00280-015-2708-9. Epub 2015 Feb 28. PMID 25724156